CLINICAL TRIAL: NCT05751863
Title: Analgesia-First Sedation in Trauma Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: MemorialCare Health System (Other)
Responsible Party: Principal Investigator, Maged Tanios, MD, Medical Director, MemorialCare Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 279-22
Record Dates: First submitted 2023-02-17; First posted 2023-03-02 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-07

CONDITIONS: Mechanical Ventilation; Respiratory Failure
Keywords: Trauma; Analgesia; Sedation; Intubation
MeSH Terms: conditions — Respiratory Insufficiency; Wounds and Injuries; Agnosia

STUDY DESIGN:
Intervention Model Description: We will enroll patients admitted into the MemorialCare Long Beach Medical Center Intensive Care Unit. Only patients admitted to the Trauma service and are mechanically ventilated, requiring continuous intravenous administration of sedatives and/or analgesics, and are anticipated to require MV for will be screened.
  Each month of the trial, the Trauma patients were assigned to use either protocol-directed sedation (PDS) plus daily sedation interruption (DSI) protocol (even numbered months) or Analgesia First Sedation (AFS) protocol (odd-numbered months). This is a pragmatic, unblinded, cluster-randomized, multiple-crossover study to evaluate the efficacy and safety of AFS versus PDS-DSI.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Analgesia First Sedation (Experimental): Subjects will be randomized to receive analgesia-first sedation by intermittent doses of Fentanyl (25 mcg), instead of continuous IV infusions. If the intermittent IVP x4 fails to achieve the target pain score, an infusion starts at 50 mcg/hr and titration by 25 mcg q15 minutes. If sedation score is not achieved, propofol infusion starts at 5 mcg/kg/min to achieve goal RASS of 0 to -2. Subjects will be assessed for a ventilator weaning trial daily.
  Interventions: Other: Analgesia First Sedation Strategy for Mechanically Ventilated (MV) Trauma Subjects
- Protocol Directed Sedation and Daily Sedation Interruption (Active Comparator): Pain management will be initiated with intravenous fentanyl at 50 mcg/hr. If the goal pain score is not achieved, use bolus doses and increase the rate by 25 mcg/hr every 15 minutes until the goal pain score is achieved. If the goal pain score is surpassed, lower the rate by 25 mcg/hr every 15 minutes. If at goal pain score, continue the current dose. If RASS scores less than the goal and Propofol is already off - decrease Fentanyl infusion.
  Agitation management will be initiated with intravenous propofol starting at 5 mcg/kg/min. Bolus doses will be used, and the rate will be increased by 5 mcg/kg/min every 15 minutes until goal RASS is achieved. If goal RASS is surpassed, lower the rate by 5 mcg/kg/min every 15 minutes until goal RASS is achieved. Bolus dose: 25 mg IVP every 5 minutes up to 2 doses PRN agitation before increasing infusion rate. Midazolam or dexmedetomidine substitutions for propofol are allowed according to the institutional protocol.
  Interventions: Other: Protocol Directed Sedation and Daily Sedation Interruption

INTERVENTIONS:
Other: Analgesia First Sedation Strategy for Mechanically Ventilated (MV) Trauma Subjects — The Intervention is using a sedation strategy for MV trauma that initially targets pain by intermittent boluses followed by an IV drip only if required. Sedatives are limited to agitation management and for a limited duration as needed. This "analgo-sedation" approach differs from the approach of using IV drips of analgesics and sedatives simultaneously and discontinuing both once daily to assess subjects.
  Arms: Analgesia First Sedation
Other: Protocol Directed Sedation and Daily Sedation Interruption — The active comparator in this study is using a sedation strategy for MV trauma that uses IV drips of analgesics and sedatives simultaneously and discontinues both once daily to assess subjects.
  Arms: Protocol Directed Sedation and Daily Sedation Interruption

SUMMARY:
The study's aim is to ascertain the best approach for providing sedation and pain management for patients who have sustained trauma and are requiring respiratory support from a mechanical ventilator. The common approach to patients who need mechanical ventilation is to provide continuous drips of sedatives and pain medicine and awaken the patient once a day to check the brain functions. Another approach is to provide pain medicine and reserve sedatives for only a short duration when needed. The difference between approaches has not been studied in Trauma patients.

DETAILED DESCRIPTION:
A significant proportion of patients admitted to the intensive care unit (ICU) require mechanical ventilation (MV). To facilitate care and maintain comfort for patients requiring MV, the utilization of a large quantity of sedatives and analgesics is required with either continuous infusion or intermittent dosing. However, prolonged continuous administration of sedatives and analgesics can contribute to prolonged MV. Numerous studies have shown that instituting protocol-directed sedation (PDS) by continuous infusion of sedatives and analgesics using a protocol that includes a daily interruption (DI) of the sedative will improve MV outcomes, specifically the duration of MV.

Protocol-directed sedation and daily sedation interruption:

Brook AD et al. performed a randomized, single-center, clinical trial; comparing protocol-directed sedation versus non-protocol-directed sedation in 321 mechanically ventilated patients. They included patients greater than the age of who were admitted to the medical intensive care unit. Based on randomization, 162 patients received protocol-directed sedation and 159 patients received non-protocol-directed sedation. The primary outcome measure was the duration of mechanical ventilation and secondary outcomes included: the length of ICU and hospital stay. The results revealed a reduction in the mean duration of mechanical ventilation for the protocol-directed sedation group (89.1 ± 133.6 hrs vs. 124.0 ± 153.6 hrs; p = .003). In addition, the protocol-directed sedation group had a reduced length of stay in the intensive care unit and hospital {5.7 ± 5.9 days vs. 7.5 ± 6.5 days (p = .013) and 14.0 ± 17.3 days vs. 19.9 ± 24.2 days (p < .001); respectively}. The protocol-directed sedation group (n = 66) had a reduced duration of continuous intravenous sedation (3.5 ± 4.0 days vs. 5.6 ± 6.4 days; p = .003). Brook's study demonstrated the clinical benefits of having protocol-directed or nurse-directed sedation in the medical intensive care unit. Since the study only involved patients in the medical intensive care unit, it is uncertain if the results are applicable to patients in the surgical unit.

Kress JP, et al. performed a randomized, single-center, clinical trial to evaluate daily interruption of continuous infusion of sedation in 128 mechanically ventilated adult patients. Notable exclusion criteria included patients already on sedative agents upon transfer to the ICU and admission due to resuscitation from cardiac arrest. The primary endpoints of the study included: the duration of mechanical ventilation, the length of stay in the intensive care unit, and the length of stay in the hospital. Total doses of sedatives (i.e. midazolam, propofol) and analgesic agents (i.e. morphine) were additional measured outcomes. Results from the study revealed a reduction in the median duration of mechanical ventilation for the daily interrupted group (4.9 vs. 7.3 days, p=.004). In addition, there was a reduction in the median length of stay in the ICU and hospital (6.4 vs. 9.9 days, p=.02 and 13.3 vs. 16.9 days, p=0.19; respectively). The total dose of midazolam was lesser in the daily interruption group (229.8 vs. 425.5 mg; p=.05). The study found no difference in regard to the incidence of self-extubation. Kress' study showed positive clinical outcomes with DI in the medical intensive care unit. However, many clinicians are concerned with the risk-related complications from DI (i.e. posttraumatic stress disorder and enhanced catecholamine response leading to cardiac complications). The study did contain limitations: it was limited to a single center and only included patients that were admitted to the medical intensive care unit. Thus, it is not clear if the results can be reproduced in other centers or applied to critically-ill surgical patients. Additionally, there was no mention of the use of PD-SBTs

Can analgesia first effectively facilitate mechanical ventilation for critically ill patients?

Strøm T et al evaluated the analgesia first in critically ill patients requiring mechanical ventilation. This was a randomized controlled trial involving 140 patients who were assigned in a 1:1 ratio to no sedation with analgesia (analgesia-first) group or sedation with DI group. The analgesia-first group or intervention arm received analgesics for pain control and sedation only if the analgesia-first approach failed. The intervention arm had significantly more days without ventilation (13.8 days ± 11.0 vs. 9.6 ± 10.0; p=0.0191) and shorter ICU days and hospital days. No difference was recorded in the occurrences of accidental extubations, but delirium was significantly higher in the analgesia-first group (20% vs. 7%, p=0.04).

Conclusion:

A literature search did not reveal any published studies demonstrating whether trauma patients should be managed with an AFS approach. This study will evaluate mechanical ventilation and ICU outcomes associated with the AFS approach to facilitate mechanical ventilation in critically ill patients. All patients will be managed with institutional-approved PDS-DSI or AFS protocols in the ICU.

- Rationale for the study

A limited number of randomized controlled trials:

Using the terms sedation and analgesia, mechanical ventilation discontinuation/weaning, critically ill, and trauma adult patients, a literature review was conducted to identify peer-reviewed articles in MEDLINE (1966-November 2021). Articles reviewed included those published in the English language, review articles, and trials with an emphasis on prospective, randomized, double-blind, placebo-controlled clinical trials. Reference citations were reviewed as an additional resource. The literature search revealed no studies that included the implementation of an AFS in trauma patients.

Which approach is preferred? There are no published studies demonstrating whether patients should be on AFS versus PDS-DSI for the management of trauma patients requiring mechanical ventilation beyond 48 hours.

How will this trial help? - Literature review

The above-mentioned literature review and search revealed no studies that included the implementation of an AFS versus PDS-DSI in ICUs. In addition, under these circumstances, it is uncertain if an AFS allowing minimal sedation is as efficacious and safe in comparison to a PDS-DSI.

- Use of trial results

The results of this study are clinically and economically relevant. The clinical data will provide information on what is the preferred sedation practice during mechanical ventilation weaning. In addition, the study will support a multi-disciplinary approach to managing mechanically ventilated patients. The measured outcomes from the study will generate further research to improve patient outcomes, specifically in mechanically ventilated patients. The economic implications can be potentially derived from the length of ICU or hospital stay.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age
2. Mechanically ventilated with an expected duration of MV ≥ 48h
3. Initiated continuous sedative/analgesic infusions by the ICU team
4. Patient is a candidate for MV weaning

Exclusion Criteria:

1. Admission after resuscitation from cardiac arrest
2. Significant neurological deficit due to a chronic disorder
3. History of alcohol dependence and/or other illicit drug abuse
4. Prior administration of continuous sedative/analgesic from a transferring institution
5. Patient receiving neuromuscular blocking agents
6. Allergy to midazolam, lorazepam, and/or propofol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2023-04-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Mechanical Ventilation days until successful extubation | 28 days
  Duration of mechanical ventilation

SECONDARY OUTCOMES:
Duration of MV weaning | 28 days
  Time from initiation of MV weaning to successful extubation

OTHER OUTCOMES:
ICU length of stay | 28 days
  Duration of ICU stay (days)
Adverse Events related to Mechanical Ventilation | 28 days
  The occurrence of any adverse event that is related to MV (e.g., unplanned extubation, delirium)

CONTACTS AND LOCATIONS:
Overall Officials: Maged Tanios, MD, MPH, Principal Investigator — Long Beach Memorial Medical Center
Locations (1):
- Long Beach Memorial Medical Center, Long Beach, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mehta S, Burry L, Cook D, Fergusson D, Steinberg M, Granton J, Herridge M, Ferguson N, Devlin J, Tanios M, Dodek P, Fowler R, Burns K, Jacka M, Olafson K, Skrobik Y, Hebert P, Sabri E, Meade M; SLEAP Investigators; Canadian Critical Care Trials Group. Daily sedation interruption in mechanically ventilated critically ill patients cared for with a sedation protocol: a randomized controlled trial. JAMA. 2012 Nov 21;308(19):1985-92. doi: 10.1001/jama.2012.13872. PMID 23180503
- [Background] Devlin JW, Skrobik Y, Gelinas C, Needham DM, Slooter AJC, Pandharipande PP, Watson PL, Weinhouse GL, Nunnally ME, Rochwerg B, Balas MC, van den Boogaard M, Bosma KJ, Brummel NE, Chanques G, Denehy L, Drouot X, Fraser GL, Harris JE, Joffe AM, Kho ME, Kress JP, Lanphere JA, McKinley S, Neufeld KJ, Pisani MA, Payen JF, Pun BT, Puntillo KA, Riker RR, Robinson BRH, Shehabi Y, Szumita PM, Winkelman C, Centofanti JE, Price C, Nikayin S, Misak CJ, Flood PD, Kiedrowski K, Alhazzani W. Clinical Practice Guidelines for the Prevention and Management of Pain, Agitation/Sedation, Delirium, Immobility, and Sleep Disruption in Adult Patients in the ICU. Crit Care Med. 2018 Sep;46(9):e825-e873. doi: 10.1097/CCM.0000000000003299. PMID 30113379
- [Background] Strom T, Martinussen T, Toft P. A protocol of no sedation for critically ill patients receiving mechanical ventilation: a randomised trial. Lancet. 2010 Feb 6;375(9713):475-80. doi: 10.1016/S0140-6736(09)62072-9. Epub 2010 Jan 29. PMID 20116842
- [Background] Kress JP, Pohlman AS, O'Connor MF, Hall JB. Daily interruption of sedative infusions in critically ill patients undergoing mechanical ventilation. N Engl J Med. 2000 May 18;342(20):1471-7. doi: 10.1056/NEJM200005183422002. PMID 10816184